CLINICAL TRIAL: NCT04622735
Title: A Comparative, Randomized, Double-blind, 3-arm Parallel, Phase III Study to Evaluate the Efficacy and Safety of a Fixed Dose Combination of Nefopam/Paracetamol Taken Orally in Moderate to Severe Pain After Impacted Third Molar Extraction
Brief Title: Nefopam/Paracetamol Fixed Dose Combination in Acute Pain After Impacted Third Molar Extraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Collaborators: Excelya (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP-CLI-2019-002
Record Dates: First submitted 2020-10-22; First posted 2020-11-10 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Pain
Keywords: Moderate to severe acute pain; Postoperative pain; Third molar extraction; Analgesics; Nefopam; Paracetamol; Multimodal analgesia; Fixed drug combination
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Nefopam; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind. Participants, investigators, and all persons involved in the conduct, data management, and analysis of the study will be fully blinded to the participant's treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FDC nefopam hydrochloride 30 mg / paracetamol 500 mg (X2) (Experimental): Each dose: 2 tablets (included in masking capsule)
  Interventions: Combination Product: nefopam hydrochloride 30mg / paracetamol 500mg X2
- Paracetamol 500 mg (X2) (Active Comparator): Each dose: 2 tablets (included in masking capsule)
  Interventions: Drug: Paracetamol 500 Mg Oral Tablet X2
- Nefopam hydrochloride 30 mg (X2) (Active Comparator): Each dose: 2 tablets (included in masking capsule)
  Interventions: Drug: Nefopam HCl 30 MG Oral Tablet X2

INTERVENTIONS:
Combination Product: nefopam hydrochloride 30mg / paracetamol 500mg X2 — The first intake is taken right after randomization. Then on-demand period (5 days maximum) respecting a 6-hour interval between intakes, and up to 3 intakes per day.
  Arms: FDC nefopam hydrochloride 30 mg / paracetamol 500 mg (X2)
Drug: Paracetamol 500 Mg Oral Tablet X2 — The first intake is taken right after randomization. Then on-demand period (5 days maximum) respecting a 6-hour interval between intakes, and up to 3 intakes per day.
  Other Names: Acetaminophen
  Arms: Paracetamol 500 mg (X2)
Drug: Nefopam HCl 30 MG Oral Tablet X2 — The first intake is taken right after randomization. Then on-demand period (5 days maximum) respecting a 6-hour interval between intakes, and up to 3 intakes per day.
  Arms: Nefopam hydrochloride 30 mg (X2)

SUMMARY:
This study aims to evaluate the analgesic efficacy of single and multiple doses of a new fixed dose combination of nefopam hydrochloride 30 mg and paracetamol 500mg taken orally in comparison to each single component.

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female patient aged from 18 years up to 65 years,
* Patient scheduled to undergo the surgical removal of at least one fully or partially impacted third mandibular molar requiring bone removal under short-acting local anaesthetic (mepivacaine or lidocaine) with or without vasoconstrictor,
* Patient weighing > 50 kg,
* Patient who has signed a written informed consent prior to any study-related procedures.

Additional inclusion criteria after surgery (randomization):

1. Patient experiencing moderate to severe pain within 4 hours after the dental extraction, defined by a baseline pain intensity Visual Analogic Scale (VAS) score ≥ 50 mm,
2. Third molar extraction(s) completed without any immediate complication, that in the opinion of the investigator, would interfere with the study conduct and/or assessments (e.g., suspected neurosensory complication, incomplete removal of tooth)

Main Exclusion Criteria:

* Patient treated by analgesics or nonsteroidal anti-inflammatory drugs (NSAIDs) within 3 days preceding the day of randomization or within 5 times the elimination half-life whichever the longest,
* Woman with positive results on a urine pregnancy test or breastfeeding woman or woman of childbearing potential without an effective contraception,
* Patient with a history of convulsive disorders,
* Patient taking mono-amine-oxidase (MAO) inhibitors (including but not limited to selegiline, isocarboxazid, tranylcypromine, phenelzine…),
* Patient with an abnormal cardiac condition: medically significant disorders of cardiac rate and/or rhythm,
* Patient with known anaemia,
* Patient with known pulmonary disease,
* Patient with known active gastric or duodenal ulcer or a history of recurrent gastrointestinal ulcer/bleeding,
* Patient with known glaucoma,
* Patients with a prostatic hyperplasia or urinary retention,
* Patient with current or chronic history of liver disease, or known hepatic or biliary abnormalities,
* Patient with a current or chronic history of severe renal impairment (glomerular filtration below 30 mL/min),

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: International Study Coordinator, Principal Investigator — Birmingham School of Dentistry
Locations (19):
- Hôpital Leuven, Leuven, Belgium
- France (5):
  - CHU Angers, Angers
  - CHU Marseille, Marseille
  - Centre Hospitalier de Pontoise, Pontoise
  - HIA Toulon, Toulon
  - CHU de tours, Tours
- Hungary (6):
  - Clinexpert Kft., Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - Swan-Med Kft., Létavértes
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház,, Nyíregyháza
  - Szent Borbála Kórház,, Tatabánya
  - Óbudai Egészségügyi Centrum, Zalaegerszeg
- Russia (3):
  - LLC Center for interdisciplinary dentistry & neuro, Moscow
  - State Medico-stomato Univ., by A.I. Evdokimov, Moscow
  - Regional clinical hospital, Yaroslavl
- United Kingdom (4):
  - Birmingham School of Dentistry, Birmingham
  - University Dental Hospital, Cardiff
  - Edinburgh Dental Institute, Edinburgh
  - BARTS HEALTH NHS TRUST Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Started | 107 | 108 | 106
Completed | 105 | 106 | 104
Not Completed | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2) | Total
Number analyzed (Participants) | 107 | 108 | 106 | 321
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 107 | 108 | 106 | 321
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (7.8) | 28.3 (7.9) | 28.3 (7.8) | 28.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 61 | 184
  Male | 45 | 47 | 45 | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 8 | 9 | 7 | 24
  Hungary | 33 | 31 | 33 | 97
  United Kingdom | 30 | 30 | 31 | 91
  France | 19 | 18 | 19 | 56
  Russia | 17 | 20 | 16 | 53

OUTCOME MEASURES:

1. Primary Outcome: Ranked Endpoints : 1. Sum of Pain Intensity Differences at 6 Hours (SPID0-6h)
Description: Pain intensity difference (PID) will be calculated using the score of pain intensity assessed by the patient at defined time points (T30, T45, T60, T90, T120, T150, T180, T240, T300, T360 min,) after the first Investigational Medicinal Product (IMP) intake and/or right before first intake of rescue medication using a 100-mm Visual Analogic Scale (VAS) compared to baseline.
  Calculation: Sum of Pain intensity difference (SPID) is the time-weighted summary measure of the total area under the pain intensity difference (PID) curve that integrates serial assessments of pain during x times after the first Investigational Medicinal Product
  SPID0-6h= SPID0-30min+SPID30min-45min+SPID45min-1h+SPID1h-1h30+SPID1h30-2h+SPID2h-2h30+SPID2h30-3h+SPID3h-4h+SPID4h-5h+SPID5h-6h With: SPIDTime1-Time2 = (PID Theoretical Time1 + PID Theoretical Time2) * (Theoretical Time2- Theoretical Time1) / 2 SPID min 0-6h = 0 SPID max 0-6h = 36000 The lower score mean a better score
Time Frame: 6 hours post-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2): Each dose: 2 tablets (included in masking capsule)
  nefopam hydrochloride 30mg / paracetamol 500mg X2: The first intake is taken right after randomization. Then on-demand period (5 days maximum) respecting a 6-hour interval between intakes, and up to 3 intakes per day.
Arm/Group | Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
score on a scale | 8955.4 (8751.8) | 8458.0 (8831.7) | 5290.7 (9109.3)
Statistical Analysis 1: Comparison: Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) vs Nefopam Hydrochloride 30 mg (X2); Test type: Superiority; p = 0.0031, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) vs Paracetamol 500 mg (X2); Test type: Superiority; p = 0.6787, Mixed Models Analysis

2. Primary Outcome: Total Pain Relief at 6 Hours (TOTPAR0-6h)
Description: Pain Relief will be assessed by the patient at defined time points (T30, T45, T60, T90, T120, T150, T180, T240, T300, T360 min) after the first IMP intake and/or right before first intake of rescue medication using a 5-point verbal rating scale (VRS).
  Calculation: TOTPAR is the time-weighted summary measure of the total area under the pain release difference curve that integrates serial assessments of pain release during x times after the first Investigational Medicinal Product TOTPAR0-6h=TOTPAR0-30min+TOTPAR30min-45min+TOTPAR45min-1h+TOTPAR1h-1h30+TOTPAR1h30-2h+TOTPAR2h-2h30+TOTPAR2h30-3h+ TOTPAR 3h-4h+ TOTPAR 4h-5h+ TOTPAR 5h-6h With: TOTPARTime1-Time2 = (PAR Time1 + PAR Time2) * (Time2-Time1) / 2 And with the score of pain relief at T0 = 0 ("none") TOTPAR min 0-6h = 0 TOTPAR max 0-6h = 1800 The higher score mean a better outcome
Time Frame: 6 hours post-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
score on a scale | 610.6 (434.5) | 602.2 (383.6) | 461.4 (384.5)

3. Primary Outcome: Proportion of Responder Patients
Description: A responder patient is a subject who achieves a reduction of 50% of pain intensity compared to baseline.
Time Frame: 6 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Participants | 47 | 43 | 35

4. Primary Outcome: The Patient's Global Impression of Change (PGIC) Questionnaire
Time Frame: 6 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 104 | 100 | 101
Participants
  VERY MUCH IMPROVED | 11 | 14 | 11
  MUCH IMPROVED | 39 | 29 | 30
  MINIMALLY IMPROVED | 22 | 24 | 31
  NO CHANGE | 14 | 12 | 13
  MINIMALLY WORSE | 10 | 12 | 7
  MUCH WORSE | 7 | 9 | 8
  VERY MUCH WORSE | 1 | 0 | 1

5. Primary Outcome: The Onset of Pain Relief
Description: Score of pain intensity will be assessed by the patient at defined time points (T30, T45, T60, T90, T120, T150, T180, T240, T300, T360 min). The time point of the first assessment obtaining a score ≤ 30 mm will be retained as time score of onset of pain relief.
Time Frame: during the first 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Participants | 76 | 74 | 58

6. Secondary Outcome: Total Pain Relief at 1 Hour (TOTPAR0-1h), 2 Hours (TOTPAR0-2h), 3 Hours (TOTPAR0-3h), and 4 Hours (TOTPAR0-4h)
Description: Pain relief (PAR) will be assessed by the patient at defined time points (T30, T45, T60, T90, T120, T150, T180, T240 min) after the first IMP intake and/or right before first intake of rescue medication using a 5-point verbal rating scale
  Calculation: TOTPAR is the time-weighted summary measure of the total area under the pain release difference curve that integrates serial assessments of pain release during x times after the first Investigational Medicinal Product TOTPAR0-6h=TOTPAR0-30min+TOTPAR30min-45min+TOTPAR45min-1h+TOTPAR1h-1h30+TOTPAR1h30-2h+TOTPAR2h-2h30+TOTPAR2h30-3h+ TOTPAR 3h-4h+ TOTPAR 4h-5h+ TOTPAR 5h-6h With: TOTPARTime1-Time2 = (PAR Time1 + PAR Time2) * (Time2-Time1) / 2 And with the score of pain relief at T0 = 0 ("none") TOTPAR min 0-any time = 0 TOTPAR max 0-1h = 300 ; TOTPAR max 0-2h = 600 ;TOTPAR max 0-3h = 900 ;TOTPAR max 0-4h = 1200 ; The higher score mean a better outcome
Time Frame: At 1 hour, 2 hours, 3 hours, and 4 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
score on a scale
  TOTPAR0-1h | 60.2 (54.2) | 69.4 (49.5) | 49.7 (47.7)
  TOTPAR0-2h | 170.0 (130.6) | 183.0 (115.7) | 133.2 (116.9)
  TOTPAR0-3h | 285.4 (210.5) | 300.8 (184.7) | 216.3 (185.7)
  TOTPAR0-4h | 399.7 (288.4) | 412.2 (252.2) | 298.4 (254.4)

7. Secondary Outcome: Sum of Pain Intensity Differences at 1 Hour (SPID0-1h), 2 Hours (SPID0-2h), 3 Hours (SPID0-3h), and 4 Hours (SPID0-4h)
Description: PID will be calculated using the score of pain intensity assessed by the patient at defined time points (T30, T45, T60, T90, T120, T150, T180, T240 min) after the first IMP intake and/or right before first intake of rescue medication using a 100-mm VAS compared to baseline.
  Calculation: SPID is the time-weighted summary measure of the total area under the pain intensity difference curve that integrates serial assessments of pain during x times after the first IMP
  SPID0-4h= SPID0-30min+SPID30min-45min+SPID45min-1h+SPID1h-1h30+SPID1h30-2h+SPID2h-2h30+SPID2h30-3h+SPID3h-4h With: SPIDTime1-Time2 = (PID Theoretical Time1 + PID Theoretical Time2) * (Theoretical Time2- Theoretical Time1) / 2 SPID min 0-any time = 0 SPID max 0-1h = 6000 ; SPID max 0-2h = 12000; SPID max 0-3h = 18000; SPID max 0-4h = 24000 The lower score mean a better score
Time Frame: At 1 hour, 2 hours, 3 hours, and 4 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
score on a scale
  SPID0-1h | 743.7 (1075.2) | 809.5 (1017.3) | 506.4 (1042.5)
  SPID0-2h | 2405.9 (2553.0) | 2418.4 (2469.2) | 1487.2 (2723.5)
  SPID0-3h | 4281.3 (4071.1) | 4128.8 (4022.0) | 2486.8 (4425.5)
  SPID0-4h | 6039.8 (5636.4) | 5786.0 (5639.1) | 3467.2 (6054.1)

8. Secondary Outcome: The Pain Intensity Differences (PID) Assessment
Description: PID will be calculated using the scores of pain intensity (VAS) at each time point compared to baseline.
  PID30min = VAS of pain intensity 30min - VAS of pain intensity baseline PID min = 0 / PID max = 100 A higher PID is a better outcome
Time Frame: At each timepoint: 30min, At 45min, until at 360 min post-dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
units on a scale
  30 min | -11.4 (22.6) | -14.8 (22.3) | -8.6 (20.8)
  45 min | -20.1 (27) | -19.6 (24.6) | -12.7 (25.9)
  360 min | -20.2 (30.2) | -18.0 (31.1) | -14.6 (29.2)

9. Secondary Outcome: Proportion of Responder Patients.
Time Frame: At 1 hour, 2 hours, 3 hours and 4 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Participants
  RESPONDER AT 1 HOUR, | 44 | 45 | 34
  RESPONDER AT 2 HOUR, | 57 | 54 | 38
  RESPONDER AT 3 HOUR, | 61 | 53 | 34
  RESPONDER AT 4 HOUR, | 54 | 50 | 37

10. Secondary Outcome: Time to the Second Investigational Medicinal Product (IMP) Intake
Time Frame: Up to 5 days after first dose
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
minutes | 438.5 [400.0 to 495.0] | 429.0 [385.0 to 480.0] | 387.0 [375.0 to 435.0]

11. Secondary Outcome: Participant Having Taken a Rescue Analgesic Treatment
Time Frame: Up to 10 days after first dose
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Participants | 19 | 26 | 35

12. Secondary Outcome: Sum of Pain Intensity Differences
Description: Pain Intensity Difference (PID) will be calculated using the score of pain intensity assessed by the patient at defined time points using a 100-mm visual Analog Scale (VAS) compared to baseline.
  Calculation: Sum of Pain Intensity Difference (SPID) is the time-weighted summary measure of the total area under the pain intensity difference curve that integrates serial assessments of pain during x times after the first Investigational Medicinal Product
  With: SPIDTime1-Time2 = (VAS Theoretical Time1 + VAS Theoretical Time2) * (Theoretical Time2- Theoretical Time1) / 2 SPID min 0-any time = 0 SPID max 0-day 1 = 144000 ; SPID max 0-day 2 = 288000 ; SPID max 0-day 3 = 432000 ; SPID max 0-day 4 = 576000 ; SPID max 0-day 5 = 720000 ; The lower score means a better outcome
Time Frame: At days 1, 2, 3, 4 and 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fixed Dose Combination Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
score on a scale
  SPID Day 1 | 23306.5 (23707.8) | 22173.7 (25105.0) | 19910.3 (28416.2)
  SPID Day 2 | 48792.4 (48167.2) | 44604.7 (48227.7) | 42972.1 (52821.9)
  SPID Day 3 | 70094.2 (70059.9) | 68351.5 (71111.0) | 61347.0 (75669.6)
  SPID Day 4 | 84261.6 (84118.3) | 84781.0 (90576.9) | 73960.7 (96674.9)
  SPID Day 5 | 92644.0 (96128.8) | 96134.2 (107774.7) | 78299.5 (106041.1)

13. Secondary Outcome: Proportion of Patients Having Taken a Rescue Analgesic Treatment Throughout the Study.
Time Frame: Up to 10 days after first dose
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Participants | 19 | 26 | 35

14. Secondary Outcome: The Total Dose of Rescue Medication Taken.
Time Frame: Up to 10 days after first dose
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 19 | 26 | 35
mg | 7.1 (5.2) | 7.3 (4.5) | 6.0 (4.0)

15. Secondary Outcome: Mean Duration Under Rescue Medication Over the 5 Days.
Time Frame: Up to 5 days after first dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 19 | 26 | 34
hours | 57.9 (51.5) | 99.4 (144.5) | 61.9 (42.2)

16. Secondary Outcome: Number of Investigational Medicinal Product (IMP) Intakes
Time Frame: Up to 5 days after first dose
Measure: Mean (Standard Deviation); unit: intake
Groups:
- Fixed Dose Combination (FDC) Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2): Each dose: 2 tablets (included in masking capsule)
  nefopam hydrochloride 30mg / paracetamol 500mg X2: The first intake is taken right after randomization. Then on-demand period (5 days maximum) respecting a 6-hour interval between intakes, and up to 3 intakes per day.
Arm/Group | Fixed Dose Combination (FDC) Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
intake | 6.4 (4.5) | 5.8 (4.2) | 5.1 (3.6)

17. Secondary Outcome: Patient's Global Impression of Change (PGIC) Score
Time Frame: Up to 10 days after first dose
Measure: Count of Participants; unit: Participants
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Participants
  VERY MUCH IMPROVED | 36 | 39 | 34
  MUCH IMPROVED | 40 | 46 | 40
  MINIMALLY IMPROVED | 11 | 9 | 16
  NO CHANGE | 9 | 4 | 5
  MINIMALLY WORSE | 3 | 1 | 1
  MUCH WORSE | 2 | 3 | 1
  VERY MUCH WORSE | 1 | 0 | 2
  Missing | 5 | 6 | 7

18. Other Pre Specified Outcome: Occurrence of Adverse Events (Serious and Non-serious Adverse Events).
Description: = Number of Events
Time Frame: Up to 10 days after first dose
Population: All population has been analysed
Measure: Number; unit: Adverse Event
Arm/Group | Fixed Dose Combination (FDC) Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
Number analyzed (Participants) | 107 | 108 | 106
Adverse Event | 39 | 25 | 35

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) | Paracetamol 500 mg (X2) | Nefopam Hydrochloride 30 mg (X2)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/108 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/108 | 0/106
Other Adverse Events (participants affected / at risk) | 39/107 | 25/108 | 35/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC Nefopam Hydrochloride 30 mg / Paracetamol 500 mg (X2) (N=107) | Paracetamol 500 mg (X2) (N=108) | Nefopam Hydrochloride 30 mg (X2) (N=106)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
MOTION SICKNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 13 (14) | 8 (8) | 13 (13)
VOMITIN (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
RETCHING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 3 (3) | 5 (5)
FATIGUE (General disorders) | 3 (3) | 2 (2) | 4 (4)
SWELLING FACE (General disorders) | 1 (1) | 2 (2) | 2 (2)
ASTHENIA (General disorders) | 1 (1) | 2 (2) | 1 (1)
CHILLS (General disorders) | 3 (3) | 1 (1) | 0 (0)
FEELING HOT (General disorders) | 0 (0) | 0 (0) | 1 (1)
ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
ALVEOLAR OSTEITIS (Infections and infestations) | 2 (3) | 3 (3) | 4 (4)
WOUND INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL OEDEMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEART RATE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TRISMUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (5) | 5 (5) | 7 (7)
DIZZINESS (Nervous system disorders) | 6 (6) | 1 (1) | 8 (8)
SOMNOLENCE (Nervous system disorders) | 7 (7) | 4 (4) | 2 (2)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
CHROMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 3 (3)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HOT FLUSH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT04622735/Prot_SAP_000.pdf